CLINICAL TRIAL: NCT00504556
Title: A Phase 2, Randomized, Parallel Group, Multi Center, Multi National Study for the Evaluation of Safety of Four Fixed Dose Regimens of DU-176b in Subjects With Non- Valvular Atrial Fibrillation
Brief Title: A Study to Assess the Safety of a Potential New Drug in Comparison to the Standard Practice of Dosing With Warfarin for Non-valvular Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DU176b-PRT018
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2015-03

CONDITIONS: Atrial Fibrillation; Thromboembolism
Keywords: Anti-coagulant; Non-valvular; Venous Thromboembolism; Prevention of Blood Clots; Atrial Fibrillation; Non-valvular atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism; Venous Thromboembolism | interventions — edoxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): DU-176b 30mg tablet once daily
  Interventions: Drug: Edoxaban (DU-176b)
- 2 (Experimental): DU-176b 60mg once daily
  Interventions: Drug: Edoxaban (DU-176b)
- 3 (Experimental): DU-176b 30mg b.i.d.
  Interventions: Drug: Edoxaban (DU-176b)
- 4 (Experimental): DU-176b 60mg tablets two times a day
  Interventions: Drug: Edoxaban (DU-176b)
- 5 (Active Comparator): warfarin tablets
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: Edoxaban (DU-176b) — 30mg tablet once daily
  Arms: 1
Drug: Edoxaban (DU-176b) — 60mg tablet once daily
  Arms: 2
Drug: Edoxaban (DU-176b) — 30mg tablet two times a day
  Arms: 3
Drug: Edoxaban (DU-176b) — 60mg tablet two times a day
  Arms: 4
Drug: warfarin — warfarin tablets
  Arms: 5

SUMMARY:
This study is to assess the safety of a potential new drug DU-176b for the prevention of stroke/systemic embolic event (SEE) in individuals with non-valvular atrial fibrillation (AF). The duration is 3 months of treatment and a 30 day follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 80 years old.
2. Able to provide written informed consent.
3. Persistent non-valvular AF supported by abnormal electrocardiogram (ECG)
4. A congestive heart failure, hypertension, age ≥ 75 years, diabetes, and prior stroke (CHADS2) index score of at least 2

Exclusion Criteria:

1. Subjects with mitral valve disease or previous valvular heart surgery
2. Known contraindication to any anticoagulant including vitamin K antagonists such as warfarin
3. Known or suspected hereditary or acquired bleeding or coagulation disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (22):
  - Huntsville, Alabama
  - Anaheim, California
  - Beverly Hills, California
  - Stockton, California
  - Orlando, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Canton, Georgia
  - Fort Wayne, Indiana
  - Iowa City, Iowa
  - Cadillac, Michigan
  - Kalispell, Montana
  - Fremont, Nebraska
  - Santa Fe, New Mexico
  - Albany, New York
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Pottstown, Pennsylvania
  - Sellersville, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
- Minsk, Belarus
- Belgium (2):
  - Brussels
  - Genk
- Bosnia and Herzegovina (4):
  - Banja Luka
  - Mostar
  - Sarajevo
  - Tuzla
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Alberta, British Columbia
  - Winnipeg, Manitoba
  - Oshawa, Ontario
  - Thunder Bay, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Chile (4):
  - Antofagasta
  - Osorno
  - Santiago
  - Temuco
- Latvia (3):
  - Daugavpils
  - Riga
  - Ventspils
- Mexico (3):
  - Córdoba
  - Guadalajara Jalisco
  - Mexico City
- Chisinau, Moldova
- Russia (24):
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Ivanovo
  - Kaliningrad
  - Kazan'
  - Kemerovo
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - N.Novgorod
  - Novosibirsk
  - Orenburg
  - Penza
  - Perm
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Saratov
  - Tomsk
  - Tula
  - Tyumen
  - Volgograd
  - Yaroslavl
- Slovakia (5):
  - Bardejov
  - Bratislava
  - Košice
  - Lučenec
  - Prešov
- Ukraine (14):
  - Cherkassy
  - Chernihiv
  - Chernivtsy
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kiev
  - Lutsk
  - Lviv
  - Odesa
  - Poltava
  - Ternopil
  - Vinnitsa
  - Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Groups:
- DU-176b 30mg qd: DU-176b 30mg tablet once daily (qd)
  Edoxaban (DU-176b): 30mg tablet once daily
- DU-176b 30mg Bid: DU-176b 30mg twice daily (bid)
  Edoxaban (DU-176b): 30mg tablet twice daily
- DU-176b 60mg qd: DU-176b 60mg once daily (qd)
  Edoxaban (DU-176b): 60mg tablet once daily
- DU-176b 60mg Bid: DU-176b 60mg tablets two times a day
  Edoxaban (DU-176b): 60mg tablet two times a day
- Warfarin Tablets: warfarin tablets
  warfarin: warfarin tablets
Period: Overall Study
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Started | 235 | 245 | 235 | 180 | 251
Safety Analysis Set | 235 | 244 | 234 | 180 | 250
Per Protocol Analysis Set | 235 | 243 | 234 | 180 | 250
Pharmacodynamic Analysis Set | 230 | 236 | 228 | 170 | 244
Completed | 200 | 207 | 204 | 52 | 226
Not Completed | 35 | 38 | 31 | 128 | 25
Not completed — Adverse Event | 11 | 11 | 14 | 13 | 5
Not completed — Death | 3 | 3 | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 3 | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 16 | 16 | 7 | 8 | 12
Not completed — administrative reasons | 0 | 2 | 2 | 1 | 2
Not completed — did not meet entry criteria | 2 | 0 | 1 | 1 | 0
Not completed — data monitor committee decision | 0 | 0 | 0 | 100 | 0
Not completed — Other | 2 | 2 | 2 | 3 | 0
Not completed — not in safety analysis set | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- DU-176b 60mg Bid: DU-176b 60mg tablet two times a day
  Edoxaban (DU-176b): 60mg tablet two times a day
- Total: Total of all reporting groups
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets | Total
Number analyzed (Participants) | 235 | 244 | 234 | 180 | 250 | 1143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 119 | 105 | 83 | 97 | 513
  >=65 years | 126 | 125 | 129 | 97 | 153 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (8.34) | 64.8 (8.83) | 64.9 (8.81) | 64.7 (8.96) | 66.0 (8.49) | 64.9 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 94 | 79 | 66 | 99 | 433
  Male | 140 | 150 | 155 | 114 | 151 | 710
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2
  White | 230 | 239 | 228 | 176 | 243 | 1116
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 5 | 4 | 7 | 23
Region of Enrollment [Number; unit: participants]
  Belarus | 5 | 5 | 6 | 1 | 5 | 22
  United States | 10 | 13 | 9 | 5 | 9 | 46
  Slovakia | 13 | 14 | 12 | 10 | 15 | 64
  Mexico | 2 | 3 | 3 | 3 | 4 | 15
  Canada | 2 | 3 | 2 | 2 | 2 | 11
  Ukraine | 77 | 80 | 81 | 70 | 83 | 391
  Russian Federation | 91 | 93 | 87 | 64 | 97 | 432
  Chile | 6 | 4 | 6 | 2 | 5 | 23
  Latvia | 5 | 6 | 6 | 4 | 6 | 27
  Moldova, Republic of | 11 | 12 | 11 | 11 | 12 | 57
  Bosnia and Herzegovina | 13 | 11 | 11 | 8 | 12 | 55

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Major Adverse Cardiac Events MACE)
Description: MACE is defined as the composite of stroke [ischemic or hemorrhagic], Systemic embolic event (SEE), Myocardial Infarction (MI), Cardiovascular (CV) death, and hospitalization for any cardiac condition
Time Frame: 3 months
Population: safety analysis set
Measure: Number (95% Confidence Interval); unit: percent of subjects experiencing events
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Number analyzed (Participants) | 235 | 244 | 234 | 180 | 250
percent of subjects experiencing events
  MACE | 1.7 [0.5 to 4.3] | 2.5 [0.9 to 5.3] | 4.3 [2.1 to 7.7] | 1.1 [0.1 to 4.0] | 2.4 [0.9 to 5.2]
  any stroke | .4 [0 to 2.3] | .8 [.1 to 2.9] | .4 [0 to 2.4] | 1.1 [0.1 to 4.0] | 1.6 [0.4 to 4.0]
  SEE | .4 [0 to 2.3] | .4 [0 to 2.3] | 0 [0 to 1.6] | 0 [0 to 2.0] | 0 [0 to 1.5]
  any stroke and/or SEE | .4 [0 to 2.3] | 1.2 [.3 to 3.6] | .4 [0 to 2.4] | 1.1 [0.1 to 4.0] | 1.6 [.4 to 4.0]
  MI | .9 [.1 to 3.0] | .4 [0 to 2.3] | .9 [.1 to 3.1] | 0 [0 to 2.0] | 0 [0 to 1.5]
  CV death | .9 [.1 to 3.0] | 1.6 [.4 to 4.1] | 0 [0 to 1.6] | 0 [0 to 2.0] | .8 [.1 to 2.9]
  hospitalization for any cardiac condition | .9 [.1 to 3.0] | .8 [.1 to 2.9] | 3.0 [1.2 to 6.1] | 0 [0 to 2.0] | .4 [0 to 2.2]

2. Primary Outcome: Adjudicated Incidence of Bleeding Events
Description: Adjudicated Incidence of Bleeding Events during treatment period
Time Frame: 3 months
Population: safety analysis set
Measure: Number (95% Confidence Interval); unit: percent of subjects with outcome event
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Number analyzed (Participants) | 235 | 244 | 234 | 180 | 250
percent of subjects with outcome event
  All bleeding | 5.5 [3.0 to 9.3] | 12.7 [8.8 to 17.5] | 7.3 [4.3 to 11.4] | 18.3 [13.0 to 24.8] | 8.0 [5.0 to 12.1]
  Major or clinically relevant non-major bleed | 3.0 [1.2 to 6.0] | 7.8 [4.8 to 11.9] | 3.8 [1.8 to 7.2] | 10.6 [6.5 to 16.0] | 3.2 [1.4 to 6.2]
  Major bleed | 0 [0 to 1.6] | 2.0 [0.7 to 4.7] | 0.4 [0 to 2.4] | 3.3 [1.2 to 7.1] | 0.4 [0 to 2.2]
Statistical Analysis 1: Comparison: DU-176b 30mg qd vs Warfarin Tablets; All bleeds; Test type: Superiority or Other; p = .367, Fisher Exact
Statistical Analysis 2: Comparison: DU-176b 30mg Bid vs Warfarin Tablets; All bleeds; Test type: Superiority or Other; p = .104, Fisher Exact
Statistical Analysis 3: Comparison: DU-176b 60mg qd vs Warfarin Tablets; All bleeds; Test type: Superiority or Other; p = .864, Fisher Exact
Statistical Analysis 4: Comparison: DU-176b 60mg Bid vs Warfarin Tablets; All bleeds; Test type: Superiority or Other; p = .002, Fisher Exact
Statistical Analysis 5: Comparison: DU-176b 30mg qd vs Warfarin Tablets; Major or Clinically Relevant (CR) non-major bleeding; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: DU-176b 30mg Bid vs Warfarin Tablets; Major or Clinically Relevant (CR) non-major bleeding; Test type: Superiority or Other; p = 0.029, Fisher Exact
Statistical Analysis 7: Comparison: DU-176b 60mg qd vs Warfarin Tablets; Major or Clinically Relevant (CR) non-major bleeding; Test type: Superiority or Other; p = 0.807, Fisher Exact
Statistical Analysis 8: Comparison: DU-176b 60mg Bid vs Warfarin Tablets; Major or Clinically Relevant (CR) non-major bleeding; Test type: Superiority or Other; p = 0.002, Fisher Exact
Statistical Analysis 9: Comparison: DU-176b 30mg qd vs Warfarin Tablets; Major bleeds; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 10: Comparison: DU-176b 30mg Bid vs Warfarin Tablets; Major bleeds; Test type: Superiority or Other; p = 0.119, Fisher Exact
Statistical Analysis 11: Comparison: DU-176b 60mg qd vs Warfarin Tablets; Major bleeds; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 12: Comparison: DU-176b 60mg Bid vs Warfarin Tablets; Major bleeds; Test type: Superiority or Other; p = 0.023, Fisher Exact

3. Secondary Outcome: Effects on Biomarker D-dimer
Description: Mean (SD) change from baseline in D-dimer
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Number analyzed (Participants) | 213 | 218 | 215 | 156 | 230
ng/mL | -225 (809.3) | -187.8 (776.8) | -100.5 (461.6) | -129.8 (771.4) | -160.7 (635.9)

4. Secondary Outcome: Effects on Biomarker Prothrombin Fragments
Description: Mean (SD) change from baseline in Prothrombin Fragments 1 and 2 (F1 and F2)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Number analyzed (Participants) | 209 | 217 | 209 | 151 | 223
pmol/L | -23.5 (1312.0) | -47.4 (1169.6) | -51.4 (868.8) | 6.4 (1353.8) | -74.6 (849.5)

5. Secondary Outcome: Pharmacokinetics (Cmin, Cmax) of DU-176b in Subjects Receiving DU-176b
Description: Median (min, max) values of Cmin,ss; Cmax,ss
Time Frame: 3 months
Measure: Median (Full Range); unit: ng/mL
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 235 | 244 | 234 | 180
ng/mL
  Cmin,ss (ng/mL) | 10.3 [3.3 to 33.8] | 21.2 [5.8 to 53.1] | 39.6 [15.4 to 71.6] | 75.7 [40.7 to 144.8]
  Cmax,ss (ng/mL) | 84.9 [48.9 to 178.8] | 173.0 [106.7 to 338.5] | 115.0 [72.9 to 240.0] | 221.4 [162.9 to 400.1]

6. Primary Outcome: Percent of Subjects With Liver-related Laboratory Marked Abnormalities (MA)
Description: liver enzyme (ALT and/or AST) and/or bilirubin (TBL) abnormalities
Time Frame: 3 months
Population: safety analysis set
Measure: Number (95% Confidence Interval); unit: percent subjects with liver related MA
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Number analyzed (Participants) | 235 | 244 | 234 | 180 | 250
percent subjects with liver related MA
  ALT, total >= 3x ULN | 1.3 [0.3 to 3.8] | 0.9 [.01 to 3.0] | 2.6 [1.0 to 5.6] | 1.7 [0.4 to 5.0] | 1.2 [0.3 to 3.5]
  AST, total >= 3x ULN | 0.9 [0.1 to 3.1] | 0.9 [0.1 to 3.0] | 1.3 [0.3 to 3.8] | 1.2 [0.1 to 4.1] | 0.8 [0.1 to 2.9]
  total bilirubin, total >= 2x ULN | 0.9 [0.1 to 3.1] | 1.3 [0.3 to 3.7] | 0.4 [0 to 2.4] | 2.9 [1.0 to 6.7] | 1.6 [0.4 to 4.1]
  ALT or AST >=3 x ULN | 1.3 [0.3 to 3.8] | 0.9 [0.1 to 3.0] | 3.1 [1.2 to 6.2] | 1.7 [0.4 to 5.0] | 1.6 [0.4 to 4.1]
  ALT or AST >=3 x ULN and TBL >=2 x ULN | 0 [0 to 1.6] | 0.4 [0 to 2.3] | 0 [0 to 1.6] | 0.6 [0 to 3.2] | 0 [0 to 1.5]

7. Secondary Outcome: Pharmacokinetics (AUC) of DU-176b in Subjects Receiving DU-176b
Description: Median (min, max) values of AUCss
Time Frame: 3 months
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 235 | 244 | 234 | 180
ng*h/mL | 825 [600 to 1862] | 1729 [1176 to 3103] | 1728 [1096 to 3125] | 3301 [2485 to 5859]

8. Secondary Outcome: Effects on Pharmacodynamic Biomarker Anti-Factor Xa Activity in Subjects Receiving DU-176b
Description: Mean (SD) change from baseline in biomarker anti-Factor Xa [FXa] activity on Day 28, 1-3 hours post dose.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 185 | 199 | 184 | 109
IU/mL | 1.46 (.96) | 1.91 (.97) | 2.42 (1.63) | 3.28 (1.46)

9. Secondary Outcome: Effects on Pharmacodynamic Biomarker (Endogenous FX Activity) in Subjects Receiving DU-176b
Description: Mean (SD) change from baseline in biomarker endogenous FX activity on Day 28, 1-3 hours post dose.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: percent change of Endogenous FX activity
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 182 | 201 | 190 | 110
percent change of Endogenous FX activity | -40.3 (26.4) | -40.2 (25.5) | -44.4 (25.7) | -45.2 (26.7)

10. Secondary Outcome: Effects on Pharmacodynamic Biomarker PICT Activity in Subjects Receiving DU-176b
Description: Mean (SD) change from baseline in biomarker prothrombinase induced clotting time [PICT] on Day 28, 1-3 hours post dose.
  PICT was determined by PICT aasay which is a plasma based functional assay to determine the anticoagulant activity on FXa and FIIa inhibition.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 181 | 196 | 180 | 110
seconds | 14.0 (5.2) | 15.4 (5.6) | 18.3 (11.9) | 19.6 (6.4)

11. Secondary Outcome: Effects on Pharmacodynamic Biomarker PT in Subjects Receiving DU-176b
Description: Mean (SD) change from baseline in biomarker prothrombin time (PT) on Day 28, 1-3 hours post dose.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 163 | 168 | 165 | 103
seconds | 0.6 (5.5) | 0.4 (6.6) | 2.0 (6.6) | 2.1 (11.7)

12. Secondary Outcome: Effects on Pharmacodynamic Biomarker INR in Subjects Receiving DU-176b
Description: Mean (SD) change from baseline in biomarker International Normalized Ratio (INR) on Day 28, 1-3 hours post dose.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid
Number analyzed (Participants) | 163 | 168 | 165 | 103
ratio | 0.05 (.51) | 0.03 (.62) | 0.17 (.61) | 0.26 (.61)

ADVERSE EVENTS:
Arm/Group | DU-176b 30mg qd | DU-176b 30mg Bid | DU-176b 60mg qd | DU-176b 60mg Bid | Warfarin Tablets
Serious Adverse Events (participants affected / at risk) | 10/235 | 16/244 | 15/234 | 14/180 | 11/250
Other Adverse Events (participants affected / at risk) | 3/235 | 8/244 | 4/234 | 10/180 | 22/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b 30mg qd (N=235) | DU-176b 30mg Bid (N=244) | DU-176b 60mg qd (N=234) | DU-176b 60mg Bid (N=180) | Warfarin Tablets (N=250)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
intestinal angina (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cerebral artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
heamorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DU-176b 30mg qd (N=235) | DU-176b 30mg Bid (N=244) | DU-176b 60mg qd (N=234) | DU-176b 60mg Bid (N=180) | Warfarin Tablets (N=250)
INR increased (Investigations) | 0 | 1 | 2 | 0 | 18
hematuria (Renal and urinary disorders) | 3 | 7 | 2 | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A study site may not publish results of a study until after a coordinated multicenter publication has been submitted for publication or until one year after the study has ended, whichever occurs first. The study site will have the opportunity to publish results of the study, provided Daiichi Sankyo has had the opportunity to review and comment on the study site's proposed publication prior to being submitted for publication with the advice of patent council and need for subject protection.